CLINICAL TRIAL: NCT01538056
Title: Physician Modified Endovascular Grafts for the Treatment of Elective, Symptomatic or Ruptured Juxtarenal Aortic Aneurysm: An Investigator Initiated Study
Brief Title: Physician Modified Endovascular Grafts
Acronym: PMEG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Benjamin W Starnes, Professor, School of Medicine: Surgery, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002977
Record Dates: First submitted 2012-02-18; First posted 2012-02-23 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Abdominal Aortic Aneurysms
Keywords: AAA
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- PMEG Fenestrated Graft or Company Manufactured Terumo Aortic Fenestrated TREO Graft (Experimental): See Interventions for more details.
  Participants who sign the informed consent form and exit the study at any timepoint will be followed via chart review for their lifespan.
  Interventions: Device: Fenestrated Endovascular Graft or Company Manufactured Terumo Aortic Fenestrated TREO Endovascular Graft

INTERVENTIONS:
Device: Fenestrated Endovascular Graft or Company Manufactured Terumo Aortic Fenestrated TREO Endovascular Graft — PMEG Fenestrated Device- Physician modified fenestrations for the bilateral renal arteries, celiac and SMA. May include several fenestrations or only one with or without the use of the Terumo Aortic TREOFit 3-D Printed Template for fenestration placement.
  Company Manufactured Device - Terumo Aortic Fenestrated TREO Abdominal Stent Graft System fenestrated for the bilateral renal arteries, celiac and SMA. May be in the straight or tapered configurations based on patient anatomical needs.
  Other Names: FEVAR

SUMMARY:
The primary objectives of this study are to determine whether physician modified endovascular grafts (PMEG) and specified company manufactured investigational devices are a safe and effective method of treating patients with elective, symptomatic or ruptured juxtarenal aortic aneurysms in those patients considered to have limited or no other options for treatment. Secondary objectives include the validation of a patient-specific, 3-D printed aortic template as a surgical planning tool for fenestrated endografting.

DETAILED DESCRIPTION:
15,000 Americans die suddenly each year from rupture of an aneurysm in the aorta, which is the ninth leading cause of death in men over age 55. Aortic aneurysms are four times more common in men than in women and usually occur in those over age 50. Approximately one percent of men between the ages of 55 and 64 will have a significant aneurysm, and the likelihood increases to about four to six percent of those men over the age of 75. In a recent population-based study of Medicare beneficiaries, 83.2% of patients undergoing endovascular repair of their aortic aneurysm were male. Furthermore, 11.9% of patients were 67 to 69 years of age, 26.8% 70 to 74, 35.7% 75 to 79, 15.8% 80 to 84 and 9.8% > 85 years of age. Ninety-six percent of patients were White, 3% Black and the rest either Hispanic or "Other". We have reason to believe that the current population of patients in the Pacific Northwest harboring abdominal aortic aneurysms match these statistics. Thus, women and minorities will definitely be under-represented in this study primarily due to the epidemiology of the disease process.

Our institution treats a large number of patients with aortic pathology including a large number of patients with symptomatic or ruptured abdominal aortic aneurysms. We recently published our results on the implementation of a protocol for managing these patients with endovascular techniques and have been able to reduce the mortality rate in half for the first time in over 30 years.

Unfortunately, not all patients presenting with symptomatic or ruptured aortic aneurysms are candidates for endovascular repair. Reasons for exclusion predominantly involve lack of a suitable proximal aortic neck. Solutions to this problem involve multi-branched or "fenestrated" endografts which are being assessed in other clinical trials. However, grafts in these trials require between 6 and 12 weeks to manufacture and deliver to the investigational site.

On-site physician modification has also been described but is currently considered outside the Instructions For Use for the intended devices. Our institution's quality improvement department recently performed an objective review of 47 consecutive PMEG cases in patients presenting with asymptomatic, symptomatic or ruptured aortic aneurysms with highly encouraging results. Many patients in our region do not have access to clinical trials involving emerging aortic endovascular therapies, and some have no other option due to urgent presentation or poor open surgical candidacy.

For these important reasons, we seek to evaluate the safety and efficacy of PMEG using FDA-approved, off-the-shelf device in order to increase the applicability of these technologies to more patients and thus save more lives. In addition, we seek to evaluate a company manufactured device, the Terumo Aortic Fenestrated TREO Stent Graft System which is very similar to the Custom-Made Fenestrated TREO that has, to date, been extensively evaluated in multiple sites throughout Europe. This device has a lower profile delivery system than other commercially available fenestrated devices and may prove to be safer and more effective than existing commercially available devices.

ELIGIBILITY:
Inclusion Criteria:

All patients must meet all of the following inclusion criteria to be eligible for enrollment into this study:

1. Patient is > 18 years of age
2. Patients who are male or non-pregnant female (females of child bearing potential must have a negative pregnancy test prior to enrollment into the study)
3. Patient or Legally Authorized Representative has signed an Institutional Review Board (IRB) approved Informed Consent Form
4. Patient has a juxtarenal abdominal aortic aneurysm that meets at least one of the following: Abdominal aortic aneurysm >5.5 cm in diameter, Aneurysm has increased in size by 0.5 cm in last 6 months, Maximum diameter of aneurysm exceeds 1.5 times the transverse dimension of an adjacent non-aneurysmal aortic segment
5. Patient has appropriate iliac/femoral artery anatomy for access, with or without the use of a conduit, that will allow endovascular access with the physician modified endovascular graft.
6. Patient has a suitable non-aneurysmal proximal aortic neck length of > 2 mm inferior to the most distal renal artery ostium.
7. Patient has a suitable non-aneurysmal distal iliac artery length (seal zone) of >15 mm. The resultant repair should preserve patency in at least one hypogastric artery.
8. Patient has a suitable non-aneurysmal proximal aortic neck diameter between 20 and 32mm, averaged across the diameters at the Celiac, SMA, at the lowest patent renal artery and at the midpoint of the renal arteries.
9. Patient has suitable non-aneurysmal distal common iliac diameters between 8 and 20 mm.
10. Patient has juxtarenal aortic neck angulation < 60º
11. Patient must be willing to comply with all required follow-up exams

Exclusion Criteria:

Patients that meet ANY of the following are not eligible for enrollment into the study:

1. Patient has a mycotic aneurysm or has an active systemic infection
2. Patient has unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina, or onset of prolonged angina)
3. Patient has a major surgical or interventional procedure planned within +/- 30 days of the AAA repair.
4. Patient has history of connective tissue disease (e.g., Marfan's or Ehler's-Danlos syndrome).
5. Patient has a known hypersensitivity or contraindication to anticoagulation or contrast media that is not amenable to pre-treatment.
6. Patient has a known allergy or intolerance stainless steel or gold
7. Patient has a body habitus that would inhibit X-ray visualization of the aorta
8. Patient has a limited life expectancy of less than 1 year
9. Patient is currently participating in another investigational device or drug clinical trial
10. Patient has other medical, social or psychological conditions that, in the opinion of the investigator, preclude them from receiving the pre-treatment, required treatment, and post-treatment procedures and evaluations.
11. Subject is eligible for enrollment in a manufacturer-sponsored IDE at the investigational site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2011-03; Primary Completion 2045-01 (Estimated); Study Completion 2055-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoints | Index Procedure through 12 Months
  The safety of physician modified endovascular grafts will be determined by evaluating the proportion of patients that experience a rate of Major Adverse Events.
Primary Effectiveness Endpoint | Index Procedure through 12 Months
  The primary effectiveness endpoint is the proportion of treatment group subjects that achieve technical and treatment success.
Primary Technical Success Endpoint | Index Procedure
  Successful delivery and deployment of the investigational device with preservation of those branch vessels intended to be preserved at the study Index Procedure.
Primary Treatment Success Endpoint | Index Procedure through 12 Months
  All the following composite endpoint criteria to be met in order for a patient to be considered a treatment success: Technical Success, Freedom from Type I & III endoleak, Freedom from stent graft migration >10mm, Freedom from AAA enlargement >5mm, Freedom from AAA rupture, Freedom from surgical conversion to open repair

SECONDARY OUTCOMES:
Secondary Safety Endpoint | Index Procedure, 12 months, End of Study, Lifespan
  The following secondary safety endpoints assessed are:, All-Cause Mortality, AAA Related Mortality, MAEs, AAA Rupture, Surgical Conversion to Open Repair.
Secondary Stent Graft Effectiveness Endpoint | Index Procedure through Lifespan
  Technical Success, Freedom from Type I & III endoleaks, Freedom from stent graft migration, Freedom from AAA enlargement >5mm.
Secondary Clinical Utility Assessment Endpoint(s) | Index Procedure
  Clinical Utility Assessment assessing overall Index Procedural items including Blood Loss, Length of Surgical Procedure, Intensive Care Unit Length of Stay, Length of Hospital Stay, and Length of Anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Starnes, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Saldana-Ruiz N, Tachida A, Mossman A, Cure R, Larimore A, Dansey K, Starnes BW, Zettervall SL. Iliac tortuosity increases reinterventions but not adverse outcomes following repair of juxtarenal aneurysms using physician-modified endografts. J Vasc Surg. 2024 Mar;79(3):497-505. doi: 10.1016/j.jvs.2023.10.053. Epub 2023 Nov 3. PMID 37923024
- [Derived] Tachida A, Stafforini N, Singh N, Starnes B, Zettervall SL. Reinterventions after physician-modified endovascular grafts for treatment of juxtarenal aortic aneurysms are non-detrimental to long-term survival. J Vasc Surg. 2023 May;77(5):1367-1374.e2. doi: 10.1016/j.jvs.2022.12.061. Epub 2023 Jan 7. PMID 36626956
- [Derived] Zettervall SL, Dansey K, Kline B, Singh N, Starnes BW. Significant aortic neck dilation occurs after repair of juxtarenal aneurysms with fenestrated endovascular aneurysm repair. J Vasc Surg. 2021 Oct;74(4):1090-1097.e2. doi: 10.1016/j.jvs.2021.03.060. Epub 2021 Apr 28. PMID 33930518
- [Derived] Hemingway JF, Starnes BW, Kline BR, Singh N. Initial experience with the Terumo aortic Treo device for fenestrated endovascular aneurysm repair. J Vasc Surg. 2021 Sep;74(3):823-831.e1. doi: 10.1016/j.jvs.2021.01.042. Epub 2021 Feb 14. PMID 33592291
- [Derived] Hurd JR, Chen X, Caps MT, Katsman D, Singh N, Zierler RE, Tatum B, Starnes BW. A reliable method for renal volume measurement and its application in fenestrated endovascular aneurysm repair. J Vasc Surg. 2020 May;71(5):1515-1520. doi: 10.1016/j.jvs.2019.07.089. Epub 2019 Oct 18. PMID 31635961
- [Derived] Starnes BW, Tatum B. Early report from an investigator-initiated investigational device exemption clinical trial on physician-modified endovascular grafts. J Vasc Surg. 2013 Aug;58(2):311-7. doi: 10.1016/j.jvs.2013.01.029. Epub 2013 May 3. PMID 23643560